CLINICAL TRIAL: NCT04227535
Title: Deciphering Rheumatoid Arthritis-associated Interstitial Lung Disease Pathogenesis 2
Acronym: TRANSLATE2
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: K170801J
Record Dates: First submitted 2019-07-15; First posted 2020-01-13 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Rheumatoid Arthritis; Interstitial Lung Disease
Keywords: Rheumatoid Arthritis; Interstitial lung disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood DNA, blood mRNA, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid arthritis - Interstitial lung disease patients: Assessment are as follows :
  1. Clinical: Demographics (e.g., age, sex, self-reported race, etc.), Health related behaviors, including smoking history, Co-morbidities and medications, Respiratory symptom assessment (e.g., cough, dyspnea), Rheumatologic assessment (e.g., disease duration, disease severity, treatment)
  2. Physiologic:Forced vital capacity (FVC), diffusing capacity for carbon monoxide (DLCO), 6-minute walk distance
  3. Radiologic: chest HRCT scan
  4. Genetic: DNA, mRNA
  5. Biologic: serum
- Rheumatoid arthritis - no Interstitial lung disease patients: Assessment are as follows :
  1. Clinical: Demographics (e.g., age, sex, self-reported race, etc.), Health related behaviors, including smoking history, Co-morbidities and medications, Respiratory symptom assessment (e.g., cough, dyspnea), Rheumatologic assessment (e.g., disease duration, disease severity, treatment)
  2. Physiologic:Forced vital capacity (FVC), diffusing capacity for carbon monoxide (DLCO), 6-minute walk distance
  3. Radiologic: chest HRCT scan
  4. Genetic: DNA, mRNA
  5. Biologic: serum

SUMMARY:
The overall goal of this study is to identify risk and prognosis factors of Interstitial Lung Disease (ILD) in patients with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
This is not an interventional study. This is a study designed to recruit individuals affected by RA and investigate associated ILD to better understand the clinical phenotypes and genetic/molecular endotypes of RAILD, including the prognosis of the disease.

ELIGIBILITY:
SELECTION OF CASES :

Inclusion Criteria:

* Age ≥18 years
* RA diagnosis according to ACR (classification of rheumatoid arthritis) 1987 and/or ACR/EULAR 2010 criteria, validated by a senior rheumatologist
* ILD diagnosis based on typical High-Resolution Computed-Tomography (HCRT) patterns and pulmonary function tests (PFT), validated by a senior pulmonologist

Exclusion Criteria:

- Lack of signed informed consent

SELECTION OF CONTROLS:

Inclusion Criteria:

* Age ≥18 years
* RA diagnosis according to ACR 1987 and/or ACR/EULAR 2010 criteria, validated by a senior rheumatologist

Exclusion Criteria:

- Lack of signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of interest are individuals affected by RA with ILD (RA-ILD). Individuals affected with RA and without ILD (RA-noILD) will be included as a control population. The ILD status being systematically assessed by HRCT chest scan.
Sampling Method: Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic factors implicated in RA-ILD using whole exome sequencing (WES). | Baseline
  whole exome sequencing data

SECONDARY OUTCOMES:
Identification of genetic factors implicated in RA-ILD using genome wide association study. | Baseline
  genome wide sequencing data
Describe RA-ILD natural history by a 5 years annual follow up of RA-ILD patients. | Every year during 5 years
  Decline of pulmonary functional tests (PFT) as well as changes in High-Resolution Computed-Tomography chest scan scores
Description of the effect of disease modifying Anti Rheumatic Drugs (DMARDs) on ILD course and mortality. | Every year during 5 years
  Influence of treatment (DMARDs and biologics) over RA-ILD course estimated annually given the cumulated dosage received.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DIEUDE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bichat Hospital, Paris, France